CLINICAL TRIAL: NCT02417818
Title: Effects of Plasma Therapy in Cutaneous Microcirculation of Different Wounds
Brief Title: Cutaneous Microcirculation After Plasma Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Kisch, MD, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-266-3
Record Dates: First submitted 2015-03-12; First posted 2015-04-16 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Burn Injury; Acute Wound; Chronic Wound; Burn Scar
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (12):
- Second-Degree Burn (Experimental): Group A (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.
  Intervention: Plasma Therapy (PlasmaDerm)
  Interventions: Device: Plasma Therapy (PlasmaDerm)
- Skin Excision (for Skin Graft) (Experimental): Group B (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of TBSA.
  Intervention: Plasma Therapy (PlasmaDerm)
  Interventions: Device: Plasma Therapy (PlasmaDerm)
- Chronic Wound (Experimental): Group C (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.
  Intervention: Plasma Therapy (PlasmaDerm)
  Interventions: Device: Plasma Therapy (PlasmaDerm)
- Intact Skin (Active Comparator): Group D (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups A-C must be evident.
  Intervention: Plasma Therapy (PlasmaDerm)
  Interventions: Device: Plasma Therapy (PlasmaDerm)
- Second-Degree Burn (repetitive) (Experimental): Group E (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.
  Intervention: Repetitive Plasma Therapy (repetitive PlasmaDerm)
  Interventions: Device: Repetitive Plasma Therapy (repetitive PlasmaDerm)
- Skin Excision (for Skin Graft) (repetitive) (Experimental): Group F (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of TBSA.
  Intervention: Repetitive Plasma Therapy (repetitive PlasmaDerm)
  Interventions: Device: Repetitive Plasma Therapy (repetitive PlasmaDerm)
- Chronic Wound (repetitive) (Experimental): Group G (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.
  Intervention: Repetitive Plasma Therapy (repetitive PlasmaDerm)
  Interventions: Device: Repetitive Plasma Therapy (repetitive PlasmaDerm)
- Intact Skin (repetitive) (Active Comparator): Group H (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups A-C must be evident.
  Intervention: Repetitive Plasma Therapy (repetitive PlasmaDerm)
  Interventions: Device: Repetitive Plasma Therapy (repetitive PlasmaDerm)
- Hypertrophic burn scar (Experimental): Group F (n=20): Consent-capable male and female patients ≥18 years of age who suffer from a hypertrophic burn scar.
  Intervention: Repetitive Plasma Therapy (repetitive PlasmaDerm)
  Interventions: Device: Plasma Therapy (PlasmaDerm)
- Hypertrophic burn scar (repetitive) (Experimental): Group F (n=20): Consent-capable male and female patients ≥18 years of age who suffer from a hypertrophic burn scar.
  Intervention: Repetitive Plasma Therapy (repetitive PlasmaDerm)
  Interventions: Device: Repetitive Plasma Therapy (repetitive PlasmaDerm)
- Flap (Experimental): Group F (n=20): Consent-capable male and female patients ≥18 years of age who received a flap.
  Intervention: Repetitive Plasma Therapy (repetitive PlasmaDerm)
  Interventions: Device: Plasma Therapy (PlasmaDerm)
- Flap (repetitive) (Experimental): Group F (n=20): Consent-capable male and female patients ≥18 years of age who received a flap.
  Intervention: Repetitive Plasma Therapy (repetitive PlasmaDerm)
  Interventions: Device: Repetitive Plasma Therapy (repetitive PlasmaDerm)

INTERVENTIONS:
Device: Plasma Therapy (PlasmaDerm) — Plasma Therapy (PlasmaDerm)
  Arms: Chronic Wound; Flap; Hypertrophic burn scar; Intact Skin; Second-Degree Burn; Skin Excision (for Skin Graft)
Device: Repetitive Plasma Therapy (repetitive PlasmaDerm) — Repetitive Plasma Therapy (Repetitive PlasmaDerm)
  Arms: Chronic Wound (repetitive); Flap (repetitive); Hypertrophic burn scar (repetitive); Intact Skin (repetitive); Second-Degree Burn (repetitive); Skin Excision (for Skin Graft) (repetitive)

SUMMARY:
In plastic and reconstructive surgery, treatment strategies of second-degree burns, superficial wounds, burn scars, flaps and chronic wounds aim at reducing infection and improving microcirculation. Although previous studies indicate that Plasma Therapy can accelerate wound healing, only a few studies focused on the elucidation of its mechanisms of action. Therefore, the aim of this study is to evaluate the microcirculatory effects of Plasma Therapy on second-degree burns, superficial wounds, burn scars, flaps and chronic wounds in a human in-vivo setting for the first time.

ELIGIBILITY:
Inclusion Criteria:

Group A (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.

Group B (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of TBSA.

Group C (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.

Group D (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups A-C must be evident. No soft tissue injury must be evident.

Group E (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.

Group F (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of TBSA.

Group G (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.

Group H (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups E-G must be evident. No soft tissue injury must be evident.

Group I (n=20): Consent-capable male and female patients ≥18 years of age suffering from a hypertrophic burn wound.

Group J (n=20): Consent-capable male and female patients ≥18 years of age suffering from a hypertrophic burn wound.

Group K (n=20): Consent-capable male and female patients ≥18 years of age received a flap.

Group L (n=20): Consent-capable male and female patients ≥18 years of age received a flap.

Exclusion Criteria:

General exclusion criteria

* below 18 years of age
* wounds requiring artificial respiration, since consent for the study participation is unobtainable

Exclusion criteria groups A, B, D, E, F, H:

* peripheral arterial occlusive disease
* vasculitis
* diabetes mellitus
* chronic kidney or liver disease
* cardiac dysfunction
* arterial hypo- or hypertension

Anamnestic exclusion criteria

* ongoing immunosuppressive or chemotherapy treatment
* drug abuse
* systemic skin diseases
* systemic and local cortisone therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Change in microcirculation (composite measure) | Baseline and 1 minute post-dose
  * capillary blood flow [arbitrary units AU]
  * capillary blood velocity [AU]
  * tissue oxygen saturation [%]
  * relative postcapillary venous filling pressure [AU]

SECONDARY OUTCOMES:
Change in microcirculation (areolar measure) | Baseline, while and 1 minute post-dose
  * tissue oxygen saturation [%]
  * tissue hemoglobin index

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Lucius J, Jensen JO, Tasar RR, Schleusser S, Stang FH, Mailander P, Kisch T. Acute Microcirculatory Effects of Remote Ischemic Conditioning in Superficial Partial Thickness Burn Wounds. J Burn Care Res. 2023 Jul 5;44(4):912-917. doi: 10.1093/jbcr/irac166. PMID 36326797